CLINICAL TRIAL: NCT06023797
Title: Retrospective Research on Lung Cancer Patients Receiving Neoadjuvant Immunochemotherapy From Zhongshan Hospital Fudan University.
Brief Title: Neoadjuvant Immunochemotherapy for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-chest
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
Keywords: neoadjuvant therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- MAICT: chemotherapy that included at one application of PD-1 inhibitor
  Interventions: Drug: Neoadjuvant immunochemotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — Patients who received NAICT and were operated at the Department of Thoracic Surgery, Zhongshan Hospital Fudan University between 2017 and 2022.
  Other Names: surgery

SUMMARY:
We retrospectively analyzed lung cancer patients who had NAICT and surgery in the Department of Thoracic Surgery, Zhongshan Hospital. NAICT was defined as chemotherapy that included at one application of PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Lung surgery was performed in the Department of Thoracic Surgery at Zhongshan Hospital;
2. At least one cycle of neoadjuvant treatment containing the immune drug PD-1 immunosuppressant was performed before surgery;
3. Malignancy was present and confirmed in the pathology before treatment and after surgery;
4. The lung lesion was the primary lesion.

Exclusion Criteria:

1. No lung surgery was performed until 2022.11;
2. No preoperative neoadjuvant therapy was performed or recorded;
3. Neoadjuvant therapy did not include immune drugs;
4. Previous history of malignancy (including surgery and adjuvant therapy);
5. Previous use of system-related immune medicines, such as immunosuppressants and monoclonal antibodies; and 6. Other conditions inappropriate for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who received NAICT and were operated at the Department of Thoracic Surgery, Zhongshan Hospital Fudan University between 2017 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2017-2023
  Progression-free defined as status of recurrence of lung cancer
Overall survival (OS) | 2017-2023
  Overall defined as the living status, alive or dead

CONTACTS AND LOCATIONS:
Locations (1):
- Zhencong Chen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided